CLINICAL TRIAL: NCT02805335
Title: Comparison Between Actually Sutureless Devices for PICC to a New Device KT FIX PLUS
Brief Title: Comparison Between Sutureless Devices for PICC and a New System KT FIX PLUS
Acronym: KTFIXPICC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A01303-44
Record Dates: First submitted 2016-03-17; First posted 2016-06-20 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Catheter Complications; Thrombosis; Displacement of Infusion Catheter; Quality of Life
Keywords: Central Venous Catheter; Catheter Bloodstream Related Infection; Economic evaluation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Group with the sutureless device actually used
- Innovative group (Experimental): Group with the new device ( KTFIX PLUS)
  Interventions: Device: KTFIX PLUS

INTERVENTIONS:
Device: KTFIX PLUS
  Arms: Innovative group

SUMMARY:
PICC (Peripherally Inserted Central Catheter) are commun used. Just one paper report morbidity with suture as fixation system for PICC (dislodgement, infection) In the guidelines it's recommended to use sutureless device. The devices actually used are unsatisfactory because of the high risk of migration, accidental removal.

A new device, called KTFIX PLUS, seem to be more secure for PICC fixation and offer the possibility to simplify the after care. This device may stay on patient for 4 weeks. Others devices may be changed 1/week.

The investigators aimed to compare morbidity between this new device and the old one. The investigators also want to perform an economic evaluation of this device and compare patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patient with indication for PICC according guidelines
* hospitalized in a departement of your hospital
* with the possibility to use a sutureless device

Exclusion Criteria:

* infection
* thrombosis
* pediatric patient
* emergency context

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
morbidity assessed as a composite of: | from baseline up to 1 year
  * Catheter infection
  * Symptomatic superficial or deep venous thrombosis
  * Catheter occlusion
  * Premature withdrawal
  * Catheter migration
  * Hematoma occurred within 24 hours after installation in incidence density

SECONDARY OUTCOMES:
quality of life | 1 year
  internal satisfaction scale
cost | 1 year
  direct costs of PICCS fastening systems
efficacy of urokinase | 1 year
  recanalization rates of PICC after application of urokinase protocol

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Fohlen, MD MSc, Principal Investigator — Medical and University Center of Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Yes